CLINICAL TRIAL: NCT05479240
Title: Neoadjuvant Chemoradiotherapy Combined With Tislelizumab in the Treatment of Locally Advanced Rectal Cancer--Randomized, Open, Multicenter Clinical Study
Brief Title: Neoadjuvant Chemoradiotherapy Combined With Tislelizumab in the Treatment of Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCO trial
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Immunotherapy
MeSH Terms: interventions — tislelizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short-range radiotherapy sequential Tislelizumab combined with chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Capecitabine; Drug: oxaliplatin; Radiation: short-range radiotherapy
- short-range radiotherapy combined with chemotherapy (Experimental)
  Interventions: Drug: Capecitabine; Drug: oxaliplatin; Radiation: short-range radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — Participants will receive Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks for 6 cycles.
  Arms: short-range radiotherapy sequential Tislelizumab combined with chemotherapy
Drug: Capecitabine — Participants will receive Capecitabine, 1000mg/m2, day 1-14 of every 3 weeks for 6 cycles
Drug: oxaliplatin — Participants will receive oxaliplatin, 130mg/m2, day 1 of every 3 weeks for 6 cycles.
Radiation: short-range radiotherapy — 5*5Gy，d1-d5

SUMMARY:
To compare the efficacy of Neoadjuvant Chemoradiotherapy Combined With/without Tislelizumab in the Treatment of Locally Advanced Rectal Cancer

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75, male or female;
* Rectal adenocarcinoma confirmed by histopathology;
* The lower margin of the tumor as assessed by MRI was below peritoneal reflex-and cT3 was associated with one or more risk factors（cT3c-d，cN1-2；MRF+；EMVI+）;
* Patients who are expected to achieve R0 resection;
* Can swallow pills normally;
* ECOG PS 0-1;
* Have not received any previous anti-tumor therapy for rectal cancer, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.;
* Surgical treatment is planned after completion of neoadjuvant therapy;
* No contraindications;
* Fertile female subjects shall have a negative serological pregnancy test within 72 hours prior to the start of trial drug administration and use effective contraceptive methods during the trial and for at least 3 months after the last dose;For male subjects with fertile female partners, effective contraceptive measures should be used during the trial period and for 3 months after the last dose;

Exclusion Criteria:

* Have a history of allergy to monoclonal antibody, tirelizumab, capecitabine, oxaliplatin or other platinum drugs;
* Have previously received or are currently receiving any of the following treatments:

A) any surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy for the tumor; B) being treated with an immunosuppressive drug or systemic hormone for immunosuppression purposes within 2 weeks prior to initial use of the study drug (dose >10mg/ day of prednisone or equivalent);In the absence of active autoimmune disease, inhaled or topical steroids and adrenocorticosteroid replacement at doses >10mg/ d of prednisone or equivalent are permitted; C) received live attenuated vaccine within 4 weeks prior to initial use of the study drug; D) major surgery or severe trauma within 4 weeks prior to first use of the study drug;

* Have any active autoimmune disease or history of autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered after hormone replacement therapy);Patients with complete remission of psoriasis or childhood asthma/allergy who do not require any intervention as adults may be considered for inclusion, but patients requiring medical intervention with bronchodilators may not be included;
* A history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation or allogeneic bone marrow transplantation;
* There is not a good control of the heart of the clinical symptoms or disease, including but not limited to: such as (1) the NYHA class II or above for heart failure, (2) the unstable angina, myocardial infarction occurred within 1 year (3), (4) have clinical significance on the chamber of sex or ventricular arrhythmias without clinical intervention or poorly controlled clinical intervention;
* Severe infection (CTCAE > level 2) occurred within 4 weeks prior to the first use of the study drug, such as severe pneumonia, bacteremia, and complications of infection requiring hospitalization;Baseline chest imaging suggests active lung inflammation, signs and symptoms of infection within 14 days prior to initial use of the study drug, or requiring oral or intravenous antibiotic treatment, except for prophylactic use of antibiotics;
* Those who were found to have active pulmonary tuberculosis infection through medical history or CT examination, or had active pulmonary tuberculosis infection history within 1 year before enrollment, or had active pulmonary tuberculosis infection history more than 1 year ago but without formal treatment;
* Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV RNA higher than the detection limit of analysis method);
* Other malignancies diagnosed within 5 years prior to the first use of the study drug, unless malignancies with a low risk of metastasis or death (5-year survival >90%), such as adequately treated basal cell carcinoma of the skin or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, may be considered for inclusion;
* Pregnant or lactating women;
* In the investigator's judgment, there are other factors that may lead to forced termination of the study, such as other serious medical conditions (including mental illness) requiring concurrent treatment, alcoholism, drug abuse, family or social factors, and factors that may affect the safety or compliance of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | 4 weeks after surgery
  Pathological examination of resected tissue samples revealed no residual tumor cells.

OTHER OUTCOMES:
Major pathological response rate | 4 weeks after surgery
  The percentage of active tumor cells in excised tissue samples was less than 10%
overall survival | every 3 months (up to 36 months）
  Defined from date of Signing ICF to date of first documentation of death from any cause or censored at the date of the last follow-up.